CLINICAL TRIAL: NCT03949738
Title: Cerebrovascular Hemodynamics and Neurocognitive Outcome in Patients With Acute Respiratory Distress Syndrome.
Brief Title: Cerebrovascular Hemodynamics in Patients With ARDS.
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: CAR ARDS
Record Dates: First submitted 2019-02-20; First posted 2019-05-14 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: ARDS
Keywords: Cerebral Autoregulation; Cerebral Hemodynamics; Cognitive Impairment; Near-infrared Spectroscopy
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with ARDS: Adults patients fulfilling the Berlin criteria for ARDS
  Interventions: Diagnostic Test: Near-infrared spectroscopy-based assessement of cerebral autoregulation.

INTERVENTIONS:
Diagnostic Test: Near-infrared spectroscopy-based assessement of cerebral autoregulation. — Cerebral autoregulation is assessed using a software that calculates correlation coefficients based on the values of cerebral oxygenation (detected by near-infrared spectroscopy) and invasively measured arterial blood pressure.
  Correlation coefficients are calculated at 10-second intervals and averaged over a period of 300 seconds, resulting in an autoregulation index (cerebral oxygenation index, COx). The index can range between -1 and +1. It provides information about cerebral autoregulation capacity, with a value below 0.3 indicating intact cerebral autoregulation.

SUMMARY:
The acute respiratory distress syndrome (ARDS) is a life-threatening disease with functional impairment of the lung. It is characterized by an excessive inflammatory response of lung tissue, capillaries, and blood vessels and is associated with high mortality. Patients who survive the acute phase of this critical disease often suffer from long-term physical, psychological, and mental sequelae, as well as persistent cognitive deficits.

In healthy individuals, autoregulatory mechanisms of the intracranial blood vessels keep blood supply to the brain independent of fluctuations in systemic blood pressure. In the case of a serious illness, these mechanisms of autoregulation may be impaired, which may favor cerebral hypoperfusion. Impairment of cerebrovascular hemodynamics can lead to neuronal damage in short and long term.

The aim of this project is to investigate cerebrovascular autoregulation in adult patients with ARDS and to evaluate the cognitive outcome at 3, 6 and 12 months after discharge from the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* ARDS

Exclusion Criteria:

* Pre-existing neurological diseases with known intracranial pathology
* Cerebrovascular disorders, including hemodynamically relevant extracranial vascular stenoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the intensive care unit of the university hospital Hamburg-Eppendorf diagnosed with ARDS.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
COx | Assessment for 60 minutes per day during the acute phase of ARDS (maximum 14 days after ARDS onset).
  Cerebral Oximetry Index (COx) as a moving correlation between arterial blood pressure and cerebral oximetry with a range from -1 to +1. A COx above 0.3 is defined as impaired cerebrovascular autoregulation. The minutes with COX above 0.3 will be assessed.

SECONDARY OUTCOMES:
Cognitive Failures Questionnaire (CFQ) | 3, 6 and 12 months after discharge from ICU.
  The Cognitive Failures Questionnaire is a self-report scale used to assess forgetfulness or inattention. It contains 25 items that are rated on a 5-point Likert scale, resulting in a total CFQ score varying from 0 to 100, with higher scores indicating more cognitive failures.
The Short Form (36) Health Survey (SF-36) | 3, 6 and 12 months after discharge from ICU.
  The SF-36 is a questionnaire used to assess patient-reported health. It contains eight health-related topics. Each topic is rated on a scale from 0 to 100 with lower scores representing more disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätskrankenhaus Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson BT, Chambers RC, Liu KD. Acute Respiratory Distress Syndrome. N Engl J Med. 2017 Aug 10;377(6):562-572. doi: 10.1056/NEJMra1608077. No abstract available. PMID 28792873
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Brown SM, Wilson EL, Presson AP, Dinglas VD, Greene T, Hopkins RO, Needham DM; with the National Institutes of Health NHLBI ARDS Network. Understanding patient outcomes after acute respiratory distress syndrome: identifying subtypes of physical, cognitive and mental health outcomes. Thorax. 2017 Dec;72(12):1094-1103. doi: 10.1136/thoraxjnl-2017-210337. Epub 2017 Aug 4. PMID 28778920
- [Background] Hopkins RO, Weaver LK, Collingridge D, Parkinson RB, Chan KJ, Orme JF Jr. Two-year cognitive, emotional, and quality-of-life outcomes in acute respiratory distress syndrome. Am J Respir Crit Care Med. 2005 Feb 15;171(4):340-7. doi: 10.1164/rccm.200406-763OC. Epub 2004 Nov 12. PMID 15542793
- [Background] Schramm P, Closhen D, Felkel M, Berres M, Klein KU, David M, Werner C, Engelhard K. Influence of PEEP on cerebral blood flow and cerebrovascular autoregulation in patients with acute respiratory distress syndrome. J Neurosurg Anesthesiol. 2013 Apr;25(2):162-7. doi: 10.1097/ANA.0b013e31827c2f46. PMID 23211642
- [Background] LASSEN NA. Cerebral blood flow and oxygen consumption in man. Physiol Rev. 1959 Apr;39(2):183-238. doi: 10.1152/physrev.1959.39.2.183. No abstract available. PMID 13645234
- [Background] Zweifel C, Dias C, Smielewski P, Czosnyka M. Continuous time-domain monitoring of cerebral autoregulation in neurocritical care. Med Eng Phys. 2014 May;36(5):638-45. doi: 10.1016/j.medengphy.2014.03.002. Epub 2014 Apr 1. PMID 24703503
- [Background] Bullinger M. [Assessment of health related quality of life with the SF-36 Health Survey]. Rehabilitation (Stuttg). 1996 Aug;35(3):XVII-XXVII; quiz XXVII-XXIX. German. PMID 8975342
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Murkin JM, Newman SP, Stump DA, Blumenthal JA. Statement of consensus on assessment of neurobehavioral outcomes after cardiac surgery. Ann Thorac Surg. 1995 May;59(5):1289-95. doi: 10.1016/0003-4975(95)00106-u. No abstract available. PMID 7733754
- [Derived] Kahl U, Yu Y, Nierhaus A, Frings D, Sensen B, Daubmann A, Kluge S, Fischer M. Cerebrovascular autoregulation and arterial carbon dioxide in patients with acute respiratory distress syndrome: a prospective observational cohort study. Ann Intensive Care. 2021 Mar 16;11(1):47. doi: 10.1186/s13613-021-00831-7. PMID 33725209